CLINICAL TRIAL: NCT03906929
Title: Exposed Versus Buried Intramedullary K-wires for Pediatric Forearm Fractures: a Randomized Controlled Trial.
Brief Title: Exposed Versus Buried Intramedullary K-wires for Pediatric Forearm Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Nabil Fouad Gergis, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: fixation of forearm fracture
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Forearm Fracture

STUDY DESIGN:
Intervention Model Description: Using of buried and exposed intramedullary k-wire in pediatric forearm fixation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pediatric forearm fracture fixed by buried or exposed intamedullary implant (Experimental): compare complication of buried or exposed intamedullary implant
  Interventions: Device: buried intramedullary K-wire; Device: exposed intramedullary K-wire

INTERVENTIONS:
Device: buried intramedullary K-wire — Using of buried kirschner wire in pediatric forearm fixation
  Other Names: buried intramedullary kirschner wire
Device: exposed intramedullary K-wire — Using of exposed kirschner wire in pediatric forearm fixation
  Other Names: exposed intramedullary kirschner wire

SUMMARY:
Comparing the rate of complications between buried and exposed intramedullary implants after fixation of pediatric forearm fractures.

DETAILED DESCRIPTION:
comparison between buried and exposed intramedullary k-wire in fixation of pediatric forearm fracture in rate of complications such as infection,malunion,nonunion and refracture.

ELIGIBILITY:
Inclusion Criteria:

1. Age: less than 10 years .
2. Diaphyseal forearm fracture.
3. closed fracture.
4. isolated or combined fracture of forearm.

Exclusion Criteria:

1. Patient age: more than 10 years old . 2-open fracture. 3- pathological fracture. 4-patient with medical history (immune compromized patient e.g D.M, cancer on chemotherapy and aplastic anemia).

5- neurovascular injury.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
compare the rate of refracture in participants who fixed by buried and exposed K-wire. | 6 months
  comparison between the rate of refractures in participants who fixed by buried and exposed K-wire by follow up every month for six month.

SECONDARY OUTCOMES:
compare the rate of infection and malunion in participants who fixed by buried and exposed K-wire. | 6 months
  compare the rate of infection and malunion in participants who fixed by buried and exposed K-wire.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Hassan, professor, Principal Investigator — professor of orthopedic and traumatology Assuit university
Locations (1):
- Assuit u. hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan LW, Siow HM. Exposed versus buried wires for fixation of lateral humeral condyle fractures in children: a comparison of safety and efficacy. J Child Orthop. 2011 Oct;5(5):329-33. doi: 10.1007/s11832-011-0358-y. Epub 2011 Jul 28. PMID 23024723
- [Background] Tsukamoto N, Mae T, Yamashita A, Hamada T, Miura T, Iguchi T, Tokunaga M, Onizuka T, Momii K, Sadashima E, Nakashima Y. Refracture of pediatric both-bone diaphyseal forearm fracture following intramedullary fixation with Kirschner wires is likely to occur in the presence of immature radiographic healing. Eur J Orthop Surg Traumatol. 2020 Oct;30(7):1231-1241. doi: 10.1007/s00590-020-02689-0. Epub 2020 May 5. PMID 32372119
- [Background] Lascombes P, Haumont T, Journeau P. Use and abuse of flexible intramedullary nailing in children and adolescents. J Pediatr Orthop. 2006 Nov-Dec;26(6):827-34. doi: 10.1097/01.bpo.0000235397.64783.d6. PMID 17065959
- [Derived] Khaled M, Fadle AA, Hassan AAA, Khalifa AA, Nabil A, Hafez A, Abol Oyoun N. To Bury or Not to Bury the K-wires After Fixation of Both Bone Forearm Fractures in Patients Younger Than 11 Years Old: A Randomized Controlled Trial. J Pediatr Orthop. 2023 Nov-Dec 01;43(10):e783-e789. doi: 10.1097/BPO.0000000000002516. Epub 2023 Sep 7. PMID 37678342